CLINICAL TRIAL: NCT02017925
Title: Pulmonary Rehabilitation in Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Pulmonary Rehabilitation in Improving Lung Function in Patients With Locally Advanced Non-Small Cell Lung Cancer Undergoing Chemoradiation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-13044; NCI-2013-02215 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Cachexia; Fatigue; Pulmonary Complications; Radiation Toxicity; Recurrent Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
Keywords: Pulmonary Rehabilitation; Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Cachexia; Fatigue; Radiation Injuries; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (early intervention) (Experimental): Beginning within 2 weeks of starting chemoradiation, patients undergo an individualized rehabilitation program comprising aerobic exercise and strength training, including treadmill walking, stationary bicycle, NU-Step, upper body resistance training and breathing retraining, 3 times per week for 8 weeks (36 sessions).
  Interventions: Behavioral: exercise intervention; Procedure: pulmonary complications management/prevention; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm II (late intervention) (Experimental): Beginning 1 month after completion of chemoradiation, patients undergo an individualized exercise rehabilitation program as in Arm I.
  Interventions: Behavioral: exercise intervention; Procedure: pulmonary complications management/prevention; Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Behavioral: exercise intervention — Undergo pulmonary rehabilitation
Procedure: pulmonary complications management/prevention — Undergo pulmonary rehabilitation
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies pulmonary rehabilitation in improving lung function in patients with locally advanced non-small cell lung cancer undergoing chemoradiation. Individualized exercise rehabilitation programs may reduce breathing problems and improve quality of life in patients with non-small cell lung cancer. It is not yet known whether pulmonary rehabilitation is more effective when started during or after cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine feasibility of pulmonary rehabilitation (PR) in patients with locally advanced unresectable non-small cell lung cancer (NSCLC) undergoing definite chemotherapy and radiation therapy.

II. To measure exercise capacity and respiratory symptoms in lung cancer patients receiving chemotherapy and radiation before and after pulmonary rehabilitation.

III. To compare if there are any differences in symptom relief, exercise capacity, and cancer treatment tolerability between performing pulmonary rehabilitation during chemo-radiation versus after completion of lung cancer treatment.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Beginning within 2 weeks of starting chemoradiation, patients undergo an individualized rehabilitation program comprising aerobic exercise and strength training, including treadmill walking, stationary bicycle, NU-Step, upper body resistance training and breathing retraining, 3 times per week for 8 weeks (36 sessions).

ARM II: Beginning 1 month after completion of chemoradiation, patients undergo an individualized exercise rehabilitation program as in Arm I.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with locally advanced unresectable NSCLC undergoing definite chemo-radiation with curative intent
* Patients must be able to sign informed consent
* Patients who qualify for pulmonary rehabilitation as part of the standard of care and are covered by medical insurance
* Patients must be able to ambulate a minimum of 100 feet prior to enrollment in pulmonary rehab
* Patients must be willing and able to travel to the pulmonary rehabilitation site at the Morehouse Medical Plaza

Exclusion Criteria:

* Tumor resection candidates
* If survival is deemed less than 6 months for any medical condition
* If they have angina or unstable coronary disease
* Congestive heart failure refractory to medical management
* Malignancy with bone instability
* Inmates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Percent improvement in the 6 minute walk from prior to post PR | Baseline to up to 8 weeks
  Either a two-sided t-test or a Wilcoxon-rank sum test will be used to test the difference in the improvement of the 6 minute walk depending on the distribution. This test will be used to compare the difference in improvement between PR during chemo-radiation of NSCLC patients and PR 8 weeks post chemo-radiation. Linear regression will be used to estimate which clinical characteristics and patient demographics are associated with improvement in 6 minute walk. The study population will be described using means and standard deviations or medians and the interquartile range.

SECONDARY OUTCOMES:
Percent improvement in the St. George Respiratory Questionnaire (SGRQ) score | Baseline to up to 8 weeks
Feasibility of the program, based on number of patients attending the sessions throughout the 8 weeks | Up to 8 weeks
  Either Pearson's chi-square of Fisher's exact methods will be used to test if the feasibility differs across groups. Logistic regression will be used to estimate which clinical characteristics and patient demographics are associated with feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Nana-Sinkam, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu